CLINICAL TRIAL: NCT06507280
Title: The Effects of Periodontal Therapy on Gingival Crevicular Fluid NLRP3,Caspase-1,IL-1β Levels in Children With Gingivitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Sultan KELES, Associate Prof. Dr., Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2024/43
Record Dates: First submitted 2024-07-02; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Gingivitis
Keywords: NLRP3; CASPASE-1; IL-1β; GINGIVITIS; GCF
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gingivitis Group (Experimental): In the first session, gingival crevicular fluid samples will be taken from teeth numbered 11,21, periodontal measurements will be made, plaques on the teeth will be cleaned and oral hygiene training will be performed. On the 7th and 30th days, gingival crevicular fluid will be taken again and periodontal measurements will be made.
  Interventions: Procedure: Periodontal theraphy
- Healthy Group (No Intervention): Gingival crevicular fluid samples will be taken from teeth numbered 11,21, periodontal measurements will be made

INTERVENTIONS:
Procedure: Periodontal theraphy — periodontal therapy
  Arms: Gingivitis Group

SUMMARY:
This study aims to determine the levels of NLRP3, caspase-1 and IL-1β concentrations in the gingival crevicular fluid of paediatric patients with gingivitis and their changes after periodontal treatment.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, necessary periodontal measurements will be performed and gingival crevicular fluid will be collected from all patients who gave written informed consent, and patients with gingivitis will be followed up on the 7th and 30th day after periodontal treatment.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the group with gingivitis;

* Systemically healthy
* 11-14 years old
* Permanent dentition
* No need for endodontic and restorative treatment
* Gingivitis with gingivitis
* Have verbally and in writing agreed to participate in the study and are willing to attend follow-up appointments regularly participants will be included in the study.

Inclusion criteria for the healthy group;

* Systemically healthy
* 11-14 years old
* Permanent dentition
* No need for endodontic and restorative treatment
* Periodontally healthy
* Have verbally and in writing agreed to participate in the study and are willing to attend follow-up appointments regularly participants will be included in the study.

Exclusion Criteria

* In need of endodontic and restorative treatment
* Systemically unhealthy
* Patients who do not give verbal or written consent

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
NLRP3 | Baseline
  NOD-, LRR- and pyrin domain-containing protein 3 level
Caspase-1 | Baseline
  Caspase-1 level
IL-1 Beta | Baseline
  Interleukin-1 Beta level

SECONDARY OUTCOMES:
NLRP3 | 7. days - 30. days
  NOD-, LRR- and pyrin domain-containing protein 3 level
Caspase-1 | 7. days -30. days
  Caspase-1 level
IL-1 Beta | 7. days-30. days
  Interleukin-1 Beta level

CONTACTS AND LOCATIONS:
Locations (1):
- Sultan Keles, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No